CLINICAL TRIAL: NCT02277392
Title: A Phase-I, Dose Escalation Study of Recombinant Human Interleukin-18 (Sb-485232) Combined With Adoptive Transfer of Vaccine-Primed CD3/CD28-Costimulated Autologous T-Cells Following Lymphodepletion for Adult Patients With Recurrent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 02814
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-07

CONDITIONS: Ovarian, Fallopian Tube and Peritoneal Cancer
MeSH Terms: interventions — Interleukin-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Vaccine---primed, CD3/CD28---costimulated autologous peripheral blood T---cells
Biological: SB---485232 (Human recombinant Interleukin---18)

SUMMARY:
This is a phase-I, dose escalation study to assess the safety and biological activity of cyclophosphamide/fludarabine lymphodepletion followed by adoptive transfer of vaccine-primed, ex vivo CD3/CD28-costimulated peripheral blood autologous T-cells, and recombinant human interleukin-18 (SB-485232, IL-18) treatment in adult patients with recurrent, Stage III or IV ovarian cancer, fallopian tube or primary peritoneal cancer who previously underwent induction vaccination with whole tumor vaccine

ELIGIBILITY:
Inclusion Criteria:

* Female greater than or equal to 18 years of age.
* Histologically confirmed diagnosis of epithelial cancer. Subject must have a measurable disease for enrollment consideration
* Subjects who have received at least one vaccine under protocol UPCC-19809 or UPCC-29810
* Predicted life expectancy of greater than or equal to 4 months.
* ECOG performance status 0 or 1.
* Must be at least 4 weeks post-operative
* No chemotherapy, immunotherapy, hormonal therapy, or biological therapy for cancer, radiotherapy, or surgical procedures (except for minor surgical procedures) within four weeks before beginning treatment with SB-485232 (six weeks for nitrosoureas and mitomycin C). Subjects must have recovered from toxicities (incurred as a result of previous therapy) sufficiently to be entered into a Phase I study.
* Blood coagulation parameters: PT such that international normalized ratio (INR) is less than or equal to 1.5 (or an in-range INR, usually between 2 and 3, if a subject is on a stable dose of therapeutic warfarin or anticoagulants for management of venous thrombosis including pulmonary thrombo-embolus) and a PTT less than 1.5 times the upper limit of normal.
* A signed and dated written informed consent form is obtained from the subject. - The subject is able to understand and comply with protocol requirements, timetables, instructions and protocol-stated restrictions.
* Normal organ and bone marrow function as defined by: - Absolute neutrophil count greater than 1,000/ul - Platelets greater than 100,000/ul - Hematocrit greater than or equal to 30 percent - AST (SGOT)/ALT(SGPT) less than 2.5 X institutional upper limit of normal - Bilirubin less than 2.0 mg/dL unless secondary to bile duct blockage by tumor - Creatinine less than1.8 mg/dL

Exclusion Criteria:

* Significant cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal or autoimmune conditions that in the opinion of the investigator places the subject at an unacceptable risk as participant in this trial.
* Subjects with any severe concurrent disease or condition, including significant active autoimmune diseases such as rheumatoid arthritis, which in the judgment of the principal investigator would make the subject inappropriate for study participation.
* Subjects who require or are likely to require more than a two-week course of corticosteroids for intercurrent illness. Subjects must complete therapy prior to enrollment. Topical corticosteroids should be stopped at least 2 weeks prior to enrollment and systemic corticosteroids should be stopped at least 4 weeks prior to enrollment.
* Subjects with any acute infection or severe or uncontrolled that requires systematic antibiotic therapy. Acute therapy must have been completed at least seven days prior to study enrollment.
* Subjects with any underlying conditions, which would contraindicate therapy with, study treatment (or allergies to reagents used in this study).
* Women who are pregnant or are breast-feeding.
* Subject has positive test result at the screening visit for one or more of the following: HTLV-1/2 and/or Anti-HIV 1 Antibody (a-HIV-1).
* Subjects receiving medications that might affect immune function. Additionally, H2 blockers are excluded, as are all antihistamines five days before and five days after each injection of study drug. NOTE: The following are exceptions: Proton pump Inhibitors (PPIs), NSAIDS including COX-2 inhibitors, acetaminophen or Enteric Coated Aspirin.
* Subjects who are positive for serum anti-Yo (cdr2) antibodies are not eligible (Yo antibody does not need to be repeated if performed in the past).
* Subjects receiving class III antiarrythmic medications.
* Subjects with any serious medical or psychiatric disorder that would interfere with subject safety or informed consent.
* Psychological,familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Known leptomeningeal disease or evidence of prior or current metastatic brain disease.
* Any investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of SB-485232.
* Subject does not have measurable disease.
* Subject has no tissue from UPCC19809 EOS biopsy and unwilling to undergo screening biopsy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States